CLINICAL TRIAL: NCT00823940
Title: A Single-blind, Randomized, Placebo Controlled, Ascending Single Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GSK1362885 in Healthy Normal Subjects.
Brief Title: A Phase 1 Study to Evaluate the Safety and Tolerability of GSK1362885 in Healthy Normal Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111497
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: FTIH; Glucagon; Safety; GSK1362885; Pharmacokinetics; Tolerability; Pharmacodynamics
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucagon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort A1 (Placebo Comparator): Dose escalation: 5 - 100mg and placebo in 4 planned doses
  Interventions: Drug: GSK1362885
- Cohort A2 (Placebo Comparator): Dose escalation: 100-600mg and placebo in 4 planned doses
  Interventions: Drug: GSK1362885
- Cohort B1 (Other): Glucagon challenge test
  Interventions: Drug: Glucagon
- Cohort B3 (Active Comparator): Glucagon challenge test + selected dose of GSK1362885
  Interventions: Drug: Glucagon + GSK1362885

INTERVENTIONS:
Drug: GSK1362885 — 5 - 100mg of GSK1362885 or placebo
  Arms: Cohort A1
Drug: GSK1362885 — 100 - 600mg or placebo
  Arms: Cohort A2
Drug: Glucagon — 0.5mg IV bolus
  Arms: Cohort B1
Drug: Glucagon + GSK1362885 — 0.5mg Glucagon IV bolus + selected dose of GSK1362885
  Arms: Cohort B3

SUMMARY:
The study will investigate whether GSK1362885 is safe and well-tolerated when administered to normal healthy subjects. The study will also measure blood levels of the study drug to determine how the body processes the drug (pharmacokinetics) and what effects the drug has on the body (pharmacodynamics).

DETAILED DESCRIPTION:
GSK1362885 is a glycogen phosphorylase inhibitor that is targeted as a treatment for Type 2 Diabetes Mellitus by reducing hepatic glucose output. This study will investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics when single doses of GSK1362885 are administered to healthy volunteers. A glucagon challenge test will be used to stimulate hepatic glucose output in order to evaluate liver glycogen phosphorylase inhibition by GSK1362885.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male or female between 18 and 55 years of age, inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea
* BMI within the range 20.0 to 31.9 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Normal cardiac function and ECG parameters, as per protocol.
* No significant rhythm abnormalities in the Screening Holter ECG recording.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of tobacco/drugs that will be screened include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks/week for men or >7 drinks/week for women.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of glycogen storage disease
* Unable or unwilling to abstain from:
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices for 7 days prior to the first dose of study medication until the final post-dose assessment at each treatment level.
* Caffeine-or xanthine-containing products for 24 hours prior to dosing until the final post-dose assessment at each treatment level.
* Use of illicit drugs
* Alcohol for 24 hours prior to dosing until final post-dose assessment at each treatment level.
* Strenuous exercise for 48 hours prior to each blood collection for clinical laboratory tests. Subjects may participate in light recreational activities during studies (e.g., watch television, read).
* History of uncorrected thyroid dysfunction or an abnormal thyroid function test assessed by TSH and free T4 at screening
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.
* History of any gastrointestinal or hepatic conditions that could impact absorption of the investigational compound.
* Significant ECG abnormalities as defined per protocol
* Resting systolic blood pressure < 80 mmHg or > 150 or diastolic blood pressure < 60 mmHg or > 90 mmHg at screening. Resting heart rate is outside the range of 45 to 100 bpm.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody.
* A positive test for HIV antibody.
* A fasting triglyceride level >400mg/dL (4.45mmol/L).
* Anemia defined by hemoglobin concentration <11.0g/dL for males or <10.0g/lL for females.
* Significant renal disease as manifested by one or more of the following:
* Creatinine clearance <80 mL/min. (estimated from serum creatinine (SCr) and demographic data using the MDRD calculation):
* Urine protein/creatinine (mg/mg) ratio >2.5; or urine albumin concentration >300 g/mg of creatinine.
* Known loss of a kidney either by surgical ablation, injury, or disease
* Subjects with values outside the specified ranges for the following key clinical laboratory tests at Screening and at readmission for each treatment period. Laboratory tests may be repeated once to confirm eligibility prior to dosing:
* Liver function tests: ALT, Direct Bilirubin, or Albumin more than 10% outside the normal reference range (<0.9 x LLN or >1.1 x ULN)
* Electrolytes: Sodium more than +/- 5mEq/L outside the normal reference range, potassium or Calcium more than 10% outside the normal reference range (<0.9 x LLN or >1.1.x ULN).
* Metabolic: Glucose more than 10% outside the normal reference range (<0.9 x LLN or >1.1 x ULN), Total Cholesterol >240mg/dl.
* Muscle: CPK >2 x ULN.
* Hematology: Hemoglobin, WBC Neutrophils, or Platelets more than 10% outside the normal reference range (<0.9 x LLN or >1.1. x ULN).
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) is prohibited from 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication until the final post-dose assessment, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Unable or unwilling to discontinue aspirin use during the study. Subjects who are taking low-dose aspirin for cardiovascular prophylaxis (81 mg or less) are eligible to participate in the study, but the aspirin must be discontinued from Screening through the Follow-up visit.

Other

* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* As a result of the medical interview, physical examination, or screening investigations, the investigator considers the subject unfit for the study.
* Subject is either an immediate family member of a participating investigator, study coordinator, employee of an investigator; or is a member of the staff conducting the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2009-01-13 (Actual); Primary Completion 2009-04-27 (Actual); Study Completion 2009-04-27 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessments including adverse events, clinical laboratory tests, electrocardiogram (ECG) and vital signs | During the duration of study participation (from 2 days up to 5 weeks)
Pharmacokinetic parameters: AUC, Cmax, Tmax, t1/2, tlag, Cl/F, and V/F | 24 - 48 hours following each dose

SECONDARY OUTCOMES:
Pharmacokinetic parameters to assess dose proportionality and food effect | 24 - 48 hours following each dose
Pharmacodynamic parameters may include change from baseline in glucose, insulin, C-peptide and AUC following administration of IV glucagon in a standardized GC test with and without prior administration of GSK1362885 | 24 - 48 hours following each dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 111497 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/111497?search=study&study_ids=111497#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 111497 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111497 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111497 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111497 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111497 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111497 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111497 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register